CLINICAL TRIAL: NCT03506373
Title: Phase II Study of Ibrutinib in Combination With Ixazomib in Patients With Waldenström Macroglobulinemia
Brief Title: Ibrutinib and Ixazomib Citrate in Treating Newly Diagnosed, Relapsed or Refractory Waldenstrom Macroglobulinemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinued after interim analysis for futility; no treatment successes observed in the first 12 patients
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC178B; NCI-2018-00595 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC178B (Other: Mayo Clinic); 18-000580 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-04-11; First posted 2018-04-24 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Waldenstrom Macroglobulinemia; Refractory Waldenstrom Macroglobulinemia; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — ibrutinib; ixazomib; Pharmacogenomic Variants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ixazomib citrate, ibrutinib) (Experimental): Patients receive ixazomib citrate PO on days 1, 8, and 15 and ibrutinib PO daily on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Ixazomib Citrate; Other: Laboratory Biomarker Analysis; Other: Pharmacodynamic Study; Other: Pharmacokinetic Study

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Drug: Ixazomib Citrate — Given PO
  Other Names: MLN-9708; MLN9708; Ninlaro
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacodynamic Study — Correlative studies
  Other Names: PHARMACODYNAMIC
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study

SUMMARY:
This phase II trial studies the side effects of ibrutinib citrate when given with ixazomib, and determines how well they work in treating patients with Waldenstrom macroglobulinemia that is newly diagnosed, has come back (recurrent) or does not respond to treatment (refractory). Enzyme inhibitors, such as ibrutinib and ixazomib citrate, may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy (as assessed by complete response [CR] rate) of the combination of ixazomib citrate (ixazomib) and ibrutinib in Waldenstrom macroglobulinemia (WM) patients.

SECONDARY OBJECTIVES:

I. To assess the overall response rate (ORR=partial response [PR] or better) in WM patients treated with ixazomib and ibrutinib.

II. To assess the time to progression (TTP) in WM patients treated with ixazomib and ibrutinib.

III. To further characterize the safety and toxicity of the combination of ibrutinib and ixazomib.

IV. To assess the overall survival (OS) in WM patients treated with ixazomib and ibrutinib.

CORRELATIVE RESEARCH OBJECTIVES:

I. To determine the role of members of the BTK signalosome in achievement or lack thereof of response to ibrutinib and ixazomib.

II. To explore biologic effects of ibrutinib and ixazomib on microenvironment in WM and correlate with response to treatment.

OUTLINE:

Patients receive ixazomib citrate orally (PO) on days 1, 8, and 15 and ibrutinib PO daily on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of WM; patients may have newly diagnosed, relapsed, or refractory disease; (definition: newly diagnosed; patients previously untreated for WM, relapse; patients who have received prior treatment for WM and now have disease recurrence; refractory; patients who have received anti-WM therapy and are noted to have progressive disease while on therapy, or those patients who demonstrated disease progression within 6 months of the last anti-WM treatment); NOTE: Ibrutinib naïve patients are allowed; if previously treated with ibrutinib, subject must have reached a response of at least stable disease (SD) and cannot have progressed while on ibrutinib; if subject stopped taking ibrutinib for reasons other than progression, they cannot have progressed for at least 6 months post last dose of ibrutinib
* Presence of measurable disease as defined by: presence of immunoglobulin M (IgM) paraprotein, measurable lymphadenopathy on imaging studies and/or physical exam, and/or bone marrow infiltration > 10%
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
* Absolute neutrophil count (ANC) >= 1000/mm^3 (obtained =< 14 days prior to registration)
* Platelet count >= 75,000/mm^3 (obtained =< 14 days prior to registration) (NOTE: platelet transfusions in order to help patients meet eligibility criteria are not allowed)
* Hemoglobin >= 9.0 g/dL (obtained =< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) unless due to Gilbert's syndrome, in which case the direct bilirubin must be =< 1.5 x ULN (obtained =< 14 days prior to registration)
* Aspartate transaminase (AST) and alanine aminotransferase (ALT) =< 3 x ULN (obtained =< 14 days prior to registration)
* Calculated creatinine clearance must be >= 30 ml/min using the Cockcroft Gault formula (obtained =< 14 days prior to registration)
* Negative pregnancy test done at screening and =< 3 days (72 hours) prior to registration, for women of childbearing potential
* Provide written informed consent
* Willingness to provide mandatory blood specimens and bone marrow specimens for correlative research
* Willingness to return to enrolling institution for follow-up

Exclusion Criteria:

* Failure to have fully recovered (i.e., =< grade 1 toxicity) from the reversible effects of prior treatment for WM
* Major surgical procedure (including open biopsy, excluding central line intravenous (IV) and port-a-cath placement) within =< 14 days prior to initiating study treatment, or anticipation of the need for major surgery during the course of the study treatment
* Radiotherapy =< 14 days prior to registration; if the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the ixazomib
* Systemic treatment, =< 14 days before registration, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or St. John's wort
* Systemic anti-cancer therapy or participation in other clinical trials, including those with other investigational agents not included in this trial, =< 28 days of registration and throughout the duration of active treatment in this trial
* Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not; prior bortezomib treatment is allowed as per: patients with prior exposure to bortezomib will be allowed if they do not have disease refractory to bortezomib)
* Central nervous system involvement (Bing-Neel syndrome)
* Infection requiring systemic antibiotic therapy or other serious infection =< 7 days prior to registration
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, serious cardiac arrhythmia requiring medication (other than adequately rate-controlled atrial fibrillation), symptomatic congestive heart failure, unstable angina, stroke/transient ischemic attack (TIA) within the past 6 months or myocardial infarction within the past 6 months
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
* Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib or ibrutinib, including difficulty swallowing
* History of any other prior malignancy; (NOTE: Exception to this are adequately treated non-melanoma skin cancers, any in situ cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for at least two years prior to study enrollment)
* Patient has >= grade 2 peripheral neuropathy or grade 1 peripheral neuropathy with pain on clinical examination during the screening period
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown

  * Pregnant women
  * Nursing women
  * Men or women of child bearing potential (WCBP) who are unwilling to employ effective contraception; effective contraception would be defined as utilizing 2 simultaneous methods of contraception from the time of signing consent through 90 days after the last dose of the study drugs unless they agree to participate in true abstinence when this is in line with the preferred and usual lifestyle of the subject; (WCBP: A female who is sexually mature and who: [1] has not undergone a hysterectomy or bilateral oophorectomy; or [2] has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time in the preceding 24 consecutive months])
* Evidence of any other serious medical condition (such as psychiatric illness, infectious diseases, physical or laboratory findings) that may interfere with the planned treatment, affect compliance or place the patient at high risk from treatment-related complications or potentially interfere with the completion of the treatment as per the protocol
* Ongoing, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive
* Liver disease with Child-Pugh class B or C liver dysfunction
* Current treatment with a combination of ibrutinib and strong CYP3A inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2025-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asher A. Chanan-Khan, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Ixazomib Citrate, Ibrutinib): Patients receive ixazomib citrate PO on days 1, 8, and 15 and ibrutinib PO daily on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.>
  > Ibrutinib: Given PO>
  > Ixazomib Citrate: Given PO>
  > Laboratory Biomarker Analysis: Correlative studies>
  > Pharmacodynamic Study: Correlative studies>
  > Pharmacokinetic Study: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Ixazomib Citrate, Ibrutinib)
Started | 21
Completed | 5
Not Completed | 16
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 2
Not completed — Disease progression | 5
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ixazomib Citrate, Ibrutinib)
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (7.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
ECOG Performance Status [Count of Participants; unit: Participants] — 0 Fully active, able to carry on all pre-disease performance without restriction>
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work>
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours>
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours>
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair>
  5. Dead
  Participants
    0 | 12
    1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CR)
Description: Complete response rate to be defined as an objective status of CR at any time, where confirmation of the complete response status is required on two consecutive evaluations with a second immunofixation before calling the patient a CR. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Categorized by Response Assessment Criteria as specified in Appendix III of the protocol.
Time Frame: 4 years
Measure: Number; unit: percentage of participants
Groups:
- Treatment (Ixazomib Citrate, Ibrutinib): Patients receive ixazomib citrate PO on days 1, 8, and 15 and ibrutinib PO daily on days 1-28. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  >
  > Ibrutinib: Given PO
  >
  > Ixazomib Citrate: Given PO
  >
  > Laboratory Biomarker Analysis: Correlative studies
  >
  > Pharmacodynamic Study: Correlative studies
  >
  > Pharmacokinetic Study: Correlative studies
Arm/Group | Treatment (Ixazomib Citrate, Ibrutinib)
Number analyzed (Participants) | 21
percentage of participants | 0

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate will be estimated by the total number of patients who achieve a CR, very good partial response (VGPR), or partial response (PR) divided by the total number of evaluable patients. All evaluable patients will be used for this analysis. Exact binomial 95% confidence intervals for the true overall response rate will be calculated. Response is categorized by Response Assessment Criteria as specified in Appendix III of the protocol.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Ixazomib Citrate, Ibrutinib)
Number analyzed (Participants) | 21
percentage of participants | 76.0 [52.83 to 91.78]

3. Secondary Outcome: Progression-free Survival
Description: The median time to progression will be estimated using the method of Kaplan-Meier. Categorized by Response Assessment Criteria as specified in Appendix III of the protocol.
Time Frame: From study registration to the earliest date of documentation of disease progression, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ixazomib Citrate, Ibrutinib)
Number analyzed (Participants) | 21
months | 22.9 [17.2 to NA] — The upper limit of the CI is not estimable due to a low number of events

4. Secondary Outcome: Overall Survival
Description: Defined as the time from study enrollment until death due to any cause. The median overall survival will be estimated using the method of Kaplan-Meier.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ixazomib Citrate, Ibrutinib)
Number analyzed (Participants) | 21
months | NA [NA to NA] — The median, upper limit and lower limit of the CI is not estimable due to a low number of events

5. Secondary Outcome: Number of Patients Experiencing Grade 3+ Adverse Effects (AE) Graded According to Common Terminology Criteria for Adverse Events (CTCAE) Version (v.) 4.0
Description: The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the AE(s) to the study treatment will be taken into consideration.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ixazomib Citrate, Ibrutinib)
Number analyzed (Participants) | 21
Participants | 13

6. Other Pre Specified Outcome: BTK Signaling Proteins (Western Blot and Densitometric Quantification) and Gene Expression (Quantitative Real-time Polymerase Chain Reaction [PCR]) Examined in CD19/CD138+ Waldenstrom Macroglobulinemia (WM) Cells
Description: 15 protein/genes associated with BTK-signaling will be assessed and their levels from baseline samples will be compared with levels from samples during treatment. Changes over time will be evaluated using paired sample approaches (Wilcoxon signed rank test). Baseline levels will be correlated with response (responder versus [vs.] non-responder) using Wilcoxon rank sum tests.
Time Frame: Up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Biologic Effects of Ibrutinib and Ixazomib Citrate on Microenvironment in WM
Description: Blood samples & bone marrow aspirate to be taken from participants. The study will explore biologic effects of ibrutinib and ixazomib on microenvironment in WM and correlate with response to treatment. Immunophenotyping of tumor infiltrating lymphocytes (TILs) using the Multi-Omyx TILs platform. This will identify 17 different types of TILs from BM samples collected at baseline and then after one cycle of treatment. This data is represented as % and actual cell counts. Next, identification of 4 types of T-cells from the blood. This will be done from peripheral blood samples collected at Baseline and then after one cycle of treatment with ixazomib + ibrutinib (Ixa+Ibr). Next, BTK receptor occupancy: This is a competitive-binding assay essentially and will be performed in CD19+/CD138+ WM cells collected at baseline and then after one cycle of treatment with Ixa+Ibr. Readout is % occupancy. Values to be correlated with response (responder vs. non-responder) using Wilcoxon rank sum tests.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Treatment (Ixazomib Citrate, Ibrutinib)
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ixazomib Citrate, Ibrutinib) (N=21)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ixazomib Citrate, Ibrutinib) (N=21)
Anemia (Blood and lymphatic system disorders) | 17 (149)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 6 (43)
Nausea (Gastrointestinal disorders) | 14 (58)
Vomiting (Gastrointestinal disorders) | 10 (21)
Edema limbs (General disorders) | 1 (2)
Fatigue (General disorders) | 16 (138)
Allergic reaction (Immune system disorders) | 1 (3)
Upper respiratory infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (4)
Platelet count decreased (Investigations) | 11 (44)
White blood cell decreased (Investigations) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Headache (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 8 (95)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (109)
Confusion (Psychiatric disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT03506373/Prot_SAP_002.pdf
  • Informed Consent Form (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03506373/ICF_001.pdf